CLINICAL TRIAL: NCT02531776
Title: Patient Experiences With Injection Needles
Acronym: NEEDLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Bente Merete Stallknecht, Professor, MD, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-6-2014-042
Record Dates: First submitted 2014-12-12; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Needle; Pen needle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subcutaneous insertions of needles (Experimental): 36 subcutaneous needle insertions per participant with 18 differently designed needles. 30test participants in total. No fluid will be injected. Pain perception will be rated by the subjects, penetration force and skin blood perfusion will be measured, and any skin reactions will be assessed.
  Interventions: Device: Subcutaneous insertions of needles

INTERVENTIONS:
Device: Subcutaneous insertions of needles — Various types of needles with different designs and mechanical properties.
  Five marketed needles are included: NovoFine 28G x 12 mm (Novo Nordisk A/S, Denmark), NovoFine 30G x 6 mm (Novo Nordisk A/S, Denmark), NovoFine 32G tip x 6 mm (Novo Nordisk A/S, Denmark), BD Ultra-Fine 32G x 4 mm Pentapoint (Beckton, Dickinson & Company, USA), and Terumo Nanopass 34G x 5 mm (Terumo, Japan).
  Ten needles have been exclusively manufactured for this clinical trial by Hart Needles, USA. These needles vary in diameter, number of needle tip grinding, and angles of grindings.
  Three needles have been modified from the original (NovoFine 32G x 6 mm) with lack of lubrication or damaged needle tip for simulations of repeated use.
  No drugs are injected. Only the needle insertion is evaluated.

SUMMARY:
This study will focus on how different injection needles are perceived by patients. The needles differ in design and mechanical properties, and will be tested in people with Type 2 Diabetes. The measured parameters during and after needle insertion are: penetration force through skin (measured with force gauge), pain perception (rated on visual analog scale, VAS, on a scale from 0 to 10), and skin blood perfusion at insertion site (measured with laser speckle contrast scanner). Furthermore, any skin reactions will be recorded.

DETAILED DESCRIPTION:
It is estimated that there presently are about 370 million diabetics in the world, and the number is increasing, particularly in newly industrialized countries, such as China and India. Approximately 90% of diabetics have Type 2 diabetes, often caused by lifestyle, such as obesity and lack of exercise. 3-5% of diabetics have Type 1 diabetes, and the cause of the disease is unknown. The remaining 5-7% have either pregnancy diabetes (temporary illness), MODY ("Maturity-Onset Diabetes of the Young") or rarer forms of diabetes.

For the treatment of Type 1 diabetes, insulin has to be injected into the subcutaneous tissue from which it is taken up into the circulation. People with Type 1 Diabetes do not produce insulin and must thus inject insulin to stabilize blood sugar levels, typically via one or two daily injections with basal insulin, as well as so-called "bolus" injections at the time of each meal. This adds up to approximately 4-5 daily insulin injections. Type 2 diabetics, who are still "early" in the disease, have reduced sensitivity to the insulin they produce, so the pancreas overproduces insulin. Beyond lifestyle changes, treatment with metformin in tablet form will in this case be the first-line drug. In the later stages of the disease, the insulin production decreases and insulin therapy should be initiated, optionally in combination with a GLP-1 analogue (Glucagon-Like Peptide-1). It is estimated that only half of all people with Type 2 diabetes are diagnosed, and that half of those diagnosed are not in treatment. Worldwide, about 27% of the treated type 2 diabetic patients receive insulin treatment, or a GLP-1 analog, 1-2 times a day.

From the above figures it can be estimated that over 100 million diabetes injections are performed globally every day. In addition, other disorders also require subcutaneous administration of drugs, e.g. growth hormone therapy or inflammatory diseases such as rheumatoid arthritis or intestinal diseases. Thus, it is of great importance that the needles used for injections, are as painless and comfortable to use as possible.

The larger needle manufacturers have for many years sought to make needles less painful and to cause less skin trauma. Until recently, these measures have primarily been making needles thinner and shorter, but now needles with alternative grindings and needle tip designs are marketed. This is to compensate for the decreased robustness of the new very thin needles, which increase the risk of the patients damaging the needle tip during an injection. Little is known, however, of how these design changes influence the perception of pain, skin damage, etc.

Despite the large market for subcutaneous needles, the methods to test newly developed needles have remained the same for many years. One of the methods frequently used is a mechanical test where the needle is passed through a rubber strip, and the penetration force is measured. This method is rapid, reproducible and with very little variation, but there are no published data comparing the force measured in the rubber strip, with that measured in humans, and how or if the penetration force in a rubber strip relates to pain, discomfort, or other physiological parameters. Smith compares the insertion forces measured in the rubber strip and in a piece of cut off porcine tissue with the conclusion that these two behave very differently and that the rubber strip is estimated to be primarily useful in testing the needle lubrication and other friction-reducing parameters.

The second method often used is a subjective patient assessment, where the test subject uses a 'Visual Analogue Scale' (VAS) to indicate how much pain he or she experiences in connection with the needle insertion. Pain indicated by VAS is a known and accepted method, but is simultaneously a measurement method with great variety, because a person's pain sensitivity depends on many things such as stress levels, emotional state, as well as expectations for the experience.

This project is innovative in that it introduces a new method for quantitatively measuring small tissue damages in the skin, as for example, a needle insertion.

The study combines technological and medical research in the form of mechanical design of medical devices and biological evaluation of mechanical impact, which in our opinion is highly relevant and quite innovative. Results from this study will be used to develop new and improved needles, which are predicted to increase patient satisfaction and make everyday life with injections easier and more convenient for the many millions of people with diabetes who every day take insulin and / or GLP-1 injections .

The method is based on the Laser Speckle technology, and measures the tissue damage in terms of the increased skin blood perfusion in connection with a needle insertion. Prior to this project, the project group performed a number of tests on pigs and the method has proven to be sensitive enough to detect differences in the blood perfusion that occurs as a result of differences in tissue damage caused by insertion of needles that vary less than 0.1 mm in diameter, Williams et al used a photoelectric pletysmografi (PPG) to investigate changes in skin blood perfusion in human subjects following injections with insulin and diluted insulin, as well as with a needle insertion to investigate the effect of the needle trauma alone. A rapid increase in blood flow was seen for all interventions. Insulin injections resulted in increased signal for more than 60 minutes after the injection, whereas the diluted liquid and the needle insertion created an increased signal for about 10 minutes. By using laser Doppler technology, Rayman et al studied how the skin circulation changed after needle insertion in people with and without diabetes. The study revealed that the people with diabetes had lower maximum-perfusion after needle insertion than the healthy subjects. Both of the above mentioned clinical studies indicate that the method obtained from the project group's pig studies could be transferred to a human study.

Thus, the study will include 35 test subjects who will receive needle insertions with 18 differently designed needles. Penetration force through the skin, pain perception and skin blood perfusion will be recorded for all needles, and any skin reactions will be recorded. By the end of the study, the following questions can be answered:

1. Which needle design parameters influence pain and skin blood perfusion, and are these two effects related?
2. Does skin blood perfusion after needle insertions in humans compare with those measured in pigs?
3. Does penetration force relate to pain and skin blood perfusion, which needle design parameters influence the force in skin, and how does it relate to the penetration force in a rubber strip?

ELIGIBILITY:
Inclusion Criteria:

Participation in the study is possible if you

* Are a man or woman with type 2 diabetes. An equal distribution of men and women is sought to compare findings between the sexes.
* Take daily injection(s) of anti-diabetic medicine (insulin or glucagon-like-peptide-1 (GLP-1) analogues) with a pen or syringe, and have done so for more than 6 months.
* Are 18-70 years (both included)
* Are slightly overweight, i.e. BMI 25-35 kg/m2.
* Are inactive for at least 6 hours before the study, i.e. transport to the investigation must be carried out without significant physical activity.
* Are Caucasian. Inclusion of other ethnicities can increase data variation and a darker skin tone can make it difficult to read any skin reactions.
* Have no significant body hair on the abdomen (can be shaved away, and if so, this should be done at least 48 hours before the test day)

Exclusion Criteria:

Participation in the study is not possible if one or more of the following criteria are met:

* Known or suspected hypersensitivity to needles, including the needle's lubricant (typically silicon oil), pen / ink color, or other materials that come into contact with the injection site
* Previous participation in the trial
* Intake of medical product which may influence pain perception within the last 14 days before trial
* Insulin pump user
* Previous surgery in the abdominal wall
* Intake of any painkillers within the last week before the test (low-dose aspirin in cardiovascular prophylactic doses is allowed)
* Known active or inactive skin diseases in the abdominal area that may influence pain perception or blood perfusion
* Anticoagulant therapy within the last month (low-dose aspirin in cardiovascular prophylactic doses is authorized, except on test day)
* Pregnant or breastfeeding
* Consumption of alcohol within the last 24 hours before the test
* Intake of drugs within the last 48 hours before the experiment
* Smokers and ex-smokers who use nicotine products (allowed if not used within the past 6 months prior to study entry)
* Moderate to severe lipodystrophy
* Severe neuropathy (grade 0/8, 1/8 or 2/8). This is examined with a Rydell-Seiffer tuning fork.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain on 0-100 mm VAS | Immediately after needle insertion.
  Pain from the needle insertions will be assessed by a 0-100 mm Visual Analog Scale where 0 mm is "no pain" and 100 mm is "worst possible pain".
Area under curve (AUC) of skin blood perfusion increase | Change from baseline (before insertion) to after insertion with continuous measurements for 15 minutes.
  Skin blood perfusion will be measured using Laser Speckle Contrast Analysis which measures the skin's perfusion in an arbitrary unit called Perfusion Units (PU). The increase in skin blood perfusion for 15 minutes after needle insertion is measured as AUC.

SECONDARY OUTCOMES:
Needle peak penetration force [N] through human skin | At time of needle insertion
  Measured with a handheld force gauge instrument, measuring the entire insertion through the skin. The peak penetration force [N] is used for comparison.
Skin reactions (bleeding, bruising, redness, swelling) on a scale from 0 to 4. | 0.5-1 hour after insertion and 20-24 hours after insertion
  The following skin reactions are evaluated and rated on a scale from 0 (no reaction) to 4 (severe reaction); bleeding, bruising, redness, and swelling. For the acute (0.5-1 hour) evaluation, the investigator evaluates the skin reactions. 20-24 hours after the subject's visit, a phone follow-up is conducted where they are asked to rate the same skin reactions for each needle insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Kezia A Præstmark, M.Sc., Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Hart JT. Rule of halves: implications of increasing diagnosis and reducing dropout for future workload and prescribing costs in primary care. Br J Gen Pract. 1992 Mar;42(356):116-9. PMID 1493028
- [Background] Smith WC, Lee AJ, Crombie IK, Tunstall-Pedoe H. Control of blood pressure in Scotland: the rule of halves. BMJ. 1990 Apr 14;300(6730):981-3. doi: 10.1136/bmj.300.6730.981. PMID 2344507
- [Background] Weinger K, Beverly EA. Barriers to achieving glycemic targets: who omits insulin and why? Diabetes Care. 2010 Feb;33(2):450-2. doi: 10.2337/dc09-2132. No abstract available. PMID 20103561
- [Background] Hirsch L, Gibney M, Berube J, Manocchio J. Impact of a modified needle tip geometry on penetration force as well as acceptability, preference, and perceived pain in subjects with diabetes. J Diabetes Sci Technol. 2012 Mar 1;6(2):328-35. doi: 10.1177/193229681200600216. PMID 22538142
- [Background] Hirsch LJ, Gibney MA, Albanese J, Qu S, Kassler-Taub K, Klaff LJ, Bailey TS. Comparative glycemic control, safety and patient ratings for a new 4 mm x 32G insulin pen needle in adults with diabetes. Curr Med Res Opin. 2010 Jun;26(6):1531-41. doi: 10.1185/03007995.2010.482499. PMID 20429832
- [Background] Jaber A, Bozzato GB, Vedrine L, Prais WA, Berube J, Laurent PE. A novel needle for subcutaneous injection of interferon beta-1a: effect on pain in volunteers and satisfaction in patients with multiple sclerosis. BMC Neurol. 2008 Oct 10;8:38. doi: 10.1186/1471-2377-8-38. PMID 18845005
- [Background] Iwanaga M, Kamoi K. Patient perceptions of injection pain and anxiety: a comparison of NovoFine 32-gauge tip 6mm and Micro Fine Plus 31-gauge 5mm needles. Diabetes Technol Ther. 2009 Feb;11(2):81-6. doi: 10.1089/dia.2008.0027. PMID 19848573
- [Background] Arendt-Nielsen L, Egekvist H, Bjerring P. Pain following controlled cutaneous insertion of needles with different diameters. Somatosens Mot Res. 2006 Mar-Jun;23(1-2):37-43. doi: 10.1080/08990220600700925. PMID 16846958
- [Background] Egekvist H, Bjerring P, Arendt-Nielsen L. Pain and mechanical injury of human skin following needle insertions. Eur J Pain. 1999 Mar;3(1):41-49. doi: 10.1053/eujp.1998.0099. PMID 10700336
- [Background] Schwartz S, Hassman D, Shelmet J, Sievers R, Weinstein R, Liang J, Lyness W. A multicenter, open-label, randomized, two-period crossover trial comparing glycemic control, satisfaction, and preference achieved with a 31 gauge x 6 mm needle versus a 29 gauge x 12.7 mm needle in obese patients with diabetes mellitus. Clin Ther. 2004 Oct;26(10):1663-78. doi: 10.1016/j.clinthera.2004.10.007. PMID 15598483
- [Background] Kreugel G, Keers JC, Kerstens MN, Wolffenbuttel BH. Randomized trial on the influence of the length of two insulin pen needles on glycemic control and patient preference in obese patients with diabetes. Diabetes Technol Ther. 2011 Jul;13(7):737-41. doi: 10.1089/dia.2011.0010. Epub 2011 Apr 10. PMID 21476936
- [Background] Praestmark KA, Jensen CB, Stallknecht B, Madsen NB, Kildegaard J. Skin blood perfusion and cellular response to insertion of insulin pen needles with different diameters. J Diabetes Sci Technol. 2014 Jul;8(4):752-9. doi: 10.1177/1932296814531099. Epub 2014 Apr 17. PMID 24876418
- [Background] Williams G, Pickup J, Clark A, Bowcock S, Cooke E, Keen H. Changes in blood flow close to subcutaneous insulin injection sites in stable and brittle diabetics. Diabetes. 1983 May;32(5):466-73. doi: 10.2337/diab.32.5.466. PMID 6341130
- [Background] Rayman G, Williams SA, Spencer PD, Smaje LH, Wise PH, Tooke JE. Impaired microvascular hyperaemic response to minor skin trauma in type I diabetes. Br Med J (Clin Res Ed). 1986 May 17;292(6531):1295-8. doi: 10.1136/bmj.292.6531.1295. PMID 2939920
- [Derived] Praestmark KA, Jensen ML, Madsen NB, Kildegaard J, Stallknecht BM. Pen needle design influences ease of insertion, pain, and skin trauma in subjects with type 2 diabetes. BMJ Open Diabetes Res Care. 2016 Dec 15;4(1):e000266. doi: 10.1136/bmjdrc-2016-000266. eCollection 2016. PMID 28074137